CLINICAL TRIAL: NCT03480139
Title: Biological Markers for the Prediction of the "Great Obstetrical Syndromes": A Longitudinal Study
Brief Title: Biomarkers in Obstetrical Complications
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999918063; 18-CH-N063
Record Dates: First submitted 2018-03-27; First posted 2018-03-29 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy; Preterm Labor; Maternal Fetal Factors; Preterm Birth
Keywords: Prematurity; Perinatal Mortality; Pregnancy Complications; Prediction of Adverse Pregnancy Outcome; Premature Rupture of Membranes; Natural History
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth; Perinatal Death; Pregnancy Complications; Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women: Pregnant women aged 18 years and older

SUMMARY:
Objective: To study the natural history of normal pregnancy and the most frequent pregnancy complications responsible for the excessive rate of perinatal morbidity and mortality, in order to develop models to predict the occurrence of these complications of pregnancy at the earliest possible time. The study focuses on the prediction of preterm labor with intact membranes, preterm prelabor rupture of membranes (PROM), preeclampsia, small for gestational age, gestational diabetes, and fetal death. These complications account for a minimum of $30 billion annually in the US alone.

Study population: A cohort of pregnant women seeking care at the prenatal clinic of the Perinatology Research Branch in Detroit, Michigan.

Design: A prospective observational cohort study of the natural history of women with a normal pregnancy, a history of adverse outcome, or those with a complication in the index pregnancy; therefore, this study will include nulliparous and parous women. Data will be collected at the time of clinic visits and will include interviews, clinical measurements, and ultrasound studies. We will assemble a biorepository of maternal biological fluids (blood, urine, saliva, cervicovaginal fluid, gingival crevicular fluid, swabs to characterize microbiota, amniotic fluid when a clinically indicated amniocentesis is performed). Placentas will be collected at the time of delivery as well as umbilical blood, and swabs to characterize the neonatal microbiota. We will use a retrospective case control and case-cohort design to generate models for the prediction of the most common pregnancy complications. These models will be developed by classifying obstetrical complications according to clinical presentation and histologic placental lesions. Models will be developed and subsequently validated in an independent cohort.

Outcome measures: The goal is to develop sensitive, specific, and parsimonious predictive models to identify the patients at risk for developing complications of pregnancy using a combination of clinical and biological markers (biochemical and biophysical).

DETAILED DESCRIPTION:
Objective: To study the natural history of normal pregnancy and the most frequent pregnancy complications responsible for the excessive rate of perinatal morbidity and mortality, in order to develop models to predict the occurrence of these complications of pregnancy at the earliest possible time. The study focuses on the prediction of preterm labor with intact membranes, preterm prelabor rupture of membranes (PROM), preeclampsia, small for gestational age, gestational diabetes, and fetal death. These complications account for a minimum of $30 billion annually in the US alone.

Study population: A cohort of pregnant women seeking care at the prenatal clinic of the Perinatology Research Branch in Detroit, Michigan.

Design: A prospective observational cohort study of the natural history of women with a normal pregnancy, a history of adverse outcome, or those with a complication in the index pregnancy; therefore, this study will include nulliparous and parous women. Data will be collected at the time of clinic visits and will include interviews, clinical measurements, and ultrasound studies. We will assemble a biorepository of maternal biological fluids (blood, urine, saliva, cervicovaginal fluid, gingival crevicular fluid, swabs to characterize microbiota, amniotic fluid when a clinically indicated amniocentesis is performed). Placentas will be collected at the time of delivery as well as umbilical blood, and swabs to characterize the neonatal microbiota. We will use a retrospective case control and case-cohort design to generate models for the prediction of the most common pregnancy complications. These models will be developed by classifying obstetrical complications according to clinical presentation and histologic placental lesions. Models will be developed and subsequently validated in an independent cohort.

Outcome measures: The goal is to develop sensitive, specific, and parsimonious predictive models to identify the patients at risk for developing complications of pregnancy using a combination of clinical and biological markers (biochemical and biophysical).

ELIGIBILITY:
* INCLUSION CRITERIA:

This prospective longitudinal cohort study will recruit consecutive pregnant women aged 18 years or more who are between 6 and 26 6/7 weeks of gestation receiving care at the Detroit Medical Center. Informed consent will be administered prior to any research procedures.

EXCLUSION CRITERIA:

Women who have high order, multiple gestations (greater than or equal to 3 fetuses) or any of the following conditions are ineligible for participation in the study: active vaginal bleeding; serious medical illness (e.g. renal insufficiency, congestive heart disease, and chronic respiratory insufficiency)

EXCLUSION CRITERIA (for MRI examination only):

* Inability to perform MRI scan due to maternal habitus
* Metallic implants that would increase risk to the patient for MRI examination
* Previous occupational exposure to metal
* History of claustrophobia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women attending Detroit Medical Center prenatal clinics in Detroit.
Sampling Method: Non-Probability Sample
Enrollment: 746 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
To develop sensitive, specific, and parsimonious predictive models to identify the patients at risk for developing complications of pregnancy using a combination of clinical and biological markers (biochemical and biophysical). | After the study is closed to accrual
  The following will be the primary outcome measures analyzed:-Preterm delivery <37, <34, and <32 weeks-Preeclampsia-Small for gestational age neonate-Fetal death-Gestational diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Wayne State University Hutzel Hospital, Detroit, Michigan, United States